CLINICAL TRIAL: NCT03509662
Title: Early High-dose Vitamin C in Post-cardiac Arrest Syndrome
Brief Title: Vitamin C in Post-cardiac Arrest
Acronym: VITaCCA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Gelderse Vallei Hospital (Other); Sint Franciscus Gasthuis (Other); Tergooiziekenhuizen (Unknown); Amphia Hospital (Other); Erasmus Medical Center (Other); Noordwest Ziekenhuisgroep (Other); Maasstad Hospital (Other); OLVG (Network)
Responsible Party: Principal Investigator, Angelique Spoelstra-de Man, M.D., Ph.D., Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL63681.029.17
Record Dates: First submitted 2018-02-15; First posted 2018-04-26 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Cardiac Arrest
Keywords: Vitamin C; Cardiac Arrest; Post-cardiac arrest syndrome; Oxidative stress
MeSH Terms: conditions — Heart Arrest; Post-Cardiac Arrest Syndrome | interventions — Ascorbic Acid; Thiamine

STUDY DESIGN:
Intervention Model Description: In this multicentre, placebo controlled double-blind randomized clinical trial patients will be recruited from the Intensive Care Units of 8 hospitals.
  270 comatose patients suffering an out-of-hospital cardiac arrest with ventricular fibrillation/tachycardia as first registered cardiac rhythm and EMV-score ≤8 will be included.
  As soon as possible patients will be randomly allocated to one of 3 treatment groups of 90 patients each and vitamin C or placebo will be started for 96 hours. Group 1 will be treated with placebo, group 2 with 2 times a day a bolus of 1.5 gr vitamin C and group 3 with 2 times a day a bolus of 5 gr vitamin C.
  All patients will receive thiamine 200 mg q 12 hourly for 4 days to limit the conversion of vitamin C to oxalate.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo group (Placebo Comparator): Group 1 will be treated with placebos for 4 days. All patients will receive Thiamine 200 mg q 12 hourly for 4 days to limit the conversion of vitamin C to oxalate
  Interventions: Drug: Thiamine; Drug: Placebos
- Vitamin C - 3 gr/day (Active Comparator): Group 2 will be treated with 1.5 gr Vitamin C b.i.d. (3 gr/day) for 4 days. All patients will receive Thiamine 200 mg q 12 hourly for 4 days to limit the conversion of vitamin C to oxalate
  Interventions: Drug: Vitamin C; Drug: Thiamine
- Vitamin C - 10 gr/day (Active Comparator): Group 3 will be treated with 5 gr Vitamin C b.i.d. (10 gr/day) for 4 days. All patients will receive Thiamine 200 mg q 12 hourly for 4 days to limit the conversion of vitamin C to oxalate
  Interventions: Drug: Vitamin C; Drug: Thiamine

INTERVENTIONS:
Drug: Vitamin C — Vitamine C will be administered intravenously as ascorbic acid (ascorbinezuur CF 100 mg/ml, Centrafarm BV, Etten Leur, Netherlands).
  Other Names: Ascorbic acid
  Arms: Vitamin C - 10 gr/day; Vitamin C - 3 gr/day
Drug: Thiamine — All patients will receive thiamine 200 mg q 12 hourly for 4 days to limit the conversion of vitamin C to oxalate.
Drug: Placebos — One group receives a placebo.
  Arms: Placebo group

SUMMARY:
Only half of the patients suffering from cardiac arrest arrive at the hospital alive. Of these survivors, more than 50% will still die or remain severely disabled. During cardiac arrest ischemia causes damage to the vital organs, especially the brain. When with return of spontaneous circulation oxygen is re-offered to the ischemic organs, massive amounts of reactive oxygen species (ROS) are produced. These ROS can further increase the damage to the myocardium and brain (reperfusion injury). Vitamin C is the primary circulating antioxidant. It scavenges free radicals and reduces the production of ROS. In a recent study we demonstrated that vitamin C plasma levels are deficient in ~60% of the patients after cardiac arrest, probably due to massive consumption. Vitamin C deficiency reduces the protection against oxidative stress. Intravenous supplementation is needed to restore deficiency and the antioxidative effect of vitamin C is much more potent if it is administered in a supraphysiological dose (≥ 3 g per day). Its strong antioxidative effect may reduce damage to the circulation and to brain, heart and other organs. Beneficial effects of high dose i.v. vitamin C after cardiac arrest have been demonstrated in preclinical studies, but not in patients.

The investigators hypothesize that vitamin C can reduce organ damage, especially cerebral injury, if administered for a short period as a high i.v. dose during the very early phase of reperfusion after cardiac arrest.

Objectives:

* To determine whether an early high dose i.v. vitamin C can improve organ function, especially neurological outcome, in patients after cardiac arrest
* To explore the optimal dosing regimen for high dose i.v. vitamin C
* To investigate in vitro the difference in effect of plasma obtained from post cardiac arrest patients treated with placebo, 3 gr/day or 10 gr/day vitamin C on endothelial cell viability and underlying oxidative pathways.

DETAILED DESCRIPTION:
Problem definition.

In Europe, each day more than 1000 patients suffer from cardiac arrest. Despite improvement of medical technologies mortality is still very high, around 75 - 80%. Of the patients who initially survive to Intensive Care Unit (ICU) admission, more than 50% still dies or remains severely disabled due to the post cardiac arrest syndrome (PCAS). Crucial in this syndrome is the overwhelming oxidative stress, which is caused by systemic ischemia/reperfusion injury and leads to destruction of endothelial function with cardiovascular failure and brain damage. Besides targeted temperature management, we have no effective therapy to improve prognosis. The levels of our primary circulating antioxidant, vitamin C, are markedly depressed after cardiac arrest. Early, high dose intravenous (iv) vitamin C administration can boost the body's antioxidant defence, and could be a new promising therapeutic intervention to improve clinical outcome by limiting oxidative damage.

Rationale high dose vitamin C.

Vitamin C administration is often wrongly considered as complementary or even alternative medicine, which does not do justice to the strong scientific base of the pleiotropic antioxidative effects of high-dose iv (not enteral!) vitamin C administration as demonstrated in multiple preclinical and clinical studies. With enteral supplementation maximally tolerated dosages cannot achieve plasma levels of > 250 µmol/l due to limited absorption. In critically ill patients, enteral supplementation even cannot restore deficiency due to the acutely increased requirements. Iv vitamin C administration generates much higher plasma levels, thus yielding more and more potent antioxidative effects. The underlying pathophysiological mechanisms are well elucidated. High plasma levels of vitamin C not only limit the generation of reactive oxygen species (ROS), repair other oxidized scavengers such as glutathione and modulate numerous enzyme reactions, but can also act as a direct radical scavenger. In addition, vitamin C maintains nitric oxide mediated endothelial integrity and vasomotor control. Furthermore, vitamin C is a cofactor in several biosynthetic pathways, such as collagen, catecholamines and peptide hormones. Deficiency will decrease there formation. Vitamin C can thereby recover endogenous vasopressor synthesis and improve wound healing.

Post cardiac arrest huge amounts of ROS are generated by various pathways. The main source of ROS are the mitochondria due to uncoupling of oxidative phosphorylation. In addition, ROS are produced by upregulated enzymes such as NADPH oxidase or during oxidation of catecholamines. When unopposed these ROS can damage virtually every biomolecule and cause severe endothelial dysfunction. This has been demonstrated in vitro: plasma derived from patients after cardiac arrest induced massive cell death of cultured endothelial cells due to pro-oxidant stress and deterioration of anti-oxidant defenses. Cell death was highest immediately after admission to the ICU.

Vitamin C depletion.

This overpowering oxidative stress during PCAS can quickly exhaust body stores of vitamin C due to massive cellular consumption and reduced regeneration. We have shown that vitamin C plasma concentrations were decreased by more than 50% compared to healthy volunteers already on the first day after cardiac arrest. After 3 days plasma concentrations further declined and more than half the patients were deficient. Low vitamin C levels were associated with multiple organ dysfunction (higher Sequential Organ Failure Assessment (SOFA) scores) and mortality. Other studies, though investigating septic and not post cardiac arrest patients, also show markedly depressed vitamin C levels on the day of admittance (~ 10 and 6 µmol/l) and an association between low vitamin C levels and multiple organ failure.

However, these deficient vitamin C levels in critically ill patients often will go unnoticed. Due to the complexity and cost of its laboratory measurement plasma levels are not available in daily practice. In addition, the vitamin C content of enteral nutrition is assumed to be sufficient. However, current nutrition protocols (even with immune enhanced nutrition) fail to normalise vitamin C levels. These low plasma levels are likely to reflect real deficiency, since they are accompanied by scorbutic intracellular leucocyte vitamin C levels as well. Even with iv vitamin C dosages up to 1 g per day vitamin C depletion persists.

(Pre) clinical studies.

Multiple preclinical experiments support the potential beneficial effect of high-dose iv vitamin C post cardiac arrest. In a rat cardiac arrest model vitamin C administration immediately after return of spontaneous circulation (ROSC) improved survival rate and neurological outcome and decreased myocardial damage. In organ-specific ischemia-reperfusion models of kidney, liver and skeletal muscle iv vitamin C ameliorated respectively renal structure and function, bile flow and cholate secretion and muscle function.

Up to now no clinical study specifically addressed the post cardiac arrest population, but several controlled studies in critically ill patients showed favourable results. In critically ill surgical patients 3 g iv vitamin C per day reduced pulmonary morbidity, new organ failure, duration of ICU/hospital stay and mortality. In burn patients very high dose iv vitamin (66 mg/kg/hr) reduced fluid requirements, body weight gain and respiratory dysfunction. In a recent pilot trial of patients with severe sepsis vitamin C both 50 mg/kg/day and 200 mg/kg/day caused earlier recovery from organ failure with reduction of the pro-inflammatory biomarkers. In a before and after study of patients with septic shock high dose iv vitamin C combined with iv thiamine and stress dose steroids substantially accelerated shock reversal and improved survival. Two studies in critically ill patients administering respectively 2.7 g/day and 1.5 g/day showed no clinical benefit. These different results might be explained by difference in timing (relatively late) and route of administration (enteral). None of the clinical studies reported negative results of vitamin C .

Safety of high dose vitamin C.

Up to now, no adverse events due to high-dose vitamin C have been reported even with extremely high dosing schedules. Theoretical risks comprise acidosis, a paradoxal pro-oxidative effect in case of iron overload, and oxalate kidney stones. In critically ill patients with sepsis 200 mg/kg/day and in cancer patients even megadoses up to 1500 mg/kg iv vitamin C three times weekly were tolerated without significant side effects. Neither these studies, nor studies in healthy volunteers reported acidosis. Vitamin C can reduce catalytic metals such as Fe2+ and Cu2+ with adverse, pro-oxidative effects in patients with hemochromatosis. These patients are excluded in most studies and will also be excluded in our study. High dose vitamin C increases urinary oxalate excretion. However, oxalate nephrocalcinosis and calcium oxalate stones take months to years to develop and none of the studies with short-term vitamin C administration reported kidney stone formation.

The investigators hypothesize that vitamin C reduces organ damage, especially cerebral injury, if administered for a short period as a high iv dose during the very early phase of reperfusion after cardiac arrest.

Primary Objective:

- To determine whether an early high dose i.v. vitamin C can improve organ function, especially neurological outcome, in patients after cardiac arrest.

Secondary Objectives:

* To explore the optimal dosing regimen for high dose i.v. vitamin C.
* To investigate in vitro the difference in effect of plasma obtained from post cardiac arrest patients treated with placebo, 3 gr/day or 10 gr/day vitamin C on endothelial cell viability and underlying oxidative pathways.

ELIGIBILITY:
Inclusion Criteria:

* An out-of-hospital cardiac arrest with return of spontaneous circulation
* Ventricular fibrillation or ventricular tachycardia as first registered cardiac rhythm
* Glasgow Coma Scale (GCS)-score ≤8.

Exclusion Criteria:

* Patients with pre-existent terminal renal insufficiency
* Known glucose 6-phosphate dehydrogenase deficiency (risk of hemolysis)
* History of urolithiasis, oxalate nephropathy or hemochromatosis
* Treatment limitations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-08-29 (Actual)

PRIMARY OUTCOMES:
The delta (Δ) Sequential Organ Failure Assessment (SOFA) score | 96 hours
  ΔSOFA score is defined as the difference between SOFA admission and SOFA at 96 hours (46). Death at 96-hours will be counted as the maximum SOFA score (24 points).

SECONDARY OUTCOMES:
Maximal Glasgow Coma Score | At 96-h and after weaning of sedation
  Neurological outcome. The Glasgow Coma Scale (GCS) is the most common scoring system used to describe the level of consciousness. The GCS measures the following functions:
  Eye opening (E): 4 = spontaneous, 3 = to sound, 2 = to pressure, 1 = none.
  Verbal response (V): 5 = orientated, 4 = confused, 3 = words, but not coherent, 2 = sounds, but no words, 1 = none.
  Motor response (M): 6 = obeys command, 5 = localizing, 4 = normal flexion, 3 = abnormal flexion, 2 = extension, 1 = none.
Cerebral Performance Categories | At 30 and 180 days
  Neurological outcome after cardiac arrest. CPC 1: Good cerebral performance (normal life) CPC 2: Moderate cerebral disability (disability but independent) CPC 3: Severe cerebral disability (conscious but disabled and dependent) CPC 4: Coma or vegetative state (unconscious) CPC 5: Brain death
Modified Rankin Scale | At 30 and 180 days
  Neurological outcome. The modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. The scale runs from 0-6, running from perfect health without symptoms to death.
  0 - No symptoms.
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. - Moderate disability. Requires some help, but able to walk unassisted.
  4. - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. - Dead.
extended Glasgow Outcome Scale | At 30 and 180 days
  Neurological outcome. The Glasgow Outcome Scale (GOS) is a global scale for functional outcome that rates patient status into one of five categories: Dead, Vegetative State, Severe Disability, Moderate Disability or Good Recovery. The Extended GOS (GOSE) provides more detailed categorization into eight categories by subdividing the categories of severe disability, moderate disability and good recovery into a lower and upper category: the scale runs from 1-8.
  1. Death
  2. Vegetative state
  3. Lower severe disability
  4. Upper severe disability
  5. Lower moderate disability
  6. Upper moderate disability
  7. Lower good recovery
  8. Upper good recovery.
HUI-3 questionnaire | At 30 and 180 days
  Neurological outcome
Neuron-specific enolase | At day 1, 2 and 3
  Neurological outcome
Intensive Care (IC)-stay | The total length of IC-stay will be determined from the date of ICU admission until the patient is discharged from the Intensive Care Unit or the date of death from any cause, assessed up to 1 year after the first day of admission.
  Clinical parameter
Hospital-stay | The total length of hospital-stay will be determined from the date of ICU admission until the patient is discharged from the hospital or the date of death from any cause assessed up to 1 year after the first day of admission.
  Clinical parameter
Mortality | 30-day
  Clinical parameter
Mortality | 180-day
  Clinical parameter
Duration of vasopressor support | When the patient is discharged from the Intensive Care or when the patient past away, the total duration of vasopressor support will be determined, assessed up to 1 year after the first day of admission.
  Clinical parameter
Troponin and CK-MB | Maximum day 1
  Myocardial injury
Lung injury score | Daily for 1 week
  Organ injury
Ventilation time | Total ventilation time during ICU stay will be determined when the patient is discharged from the ICU or when the patient past away from any cause, assessed up to 1 year after the first day of admission.
Renal function | eGFR will be measured daily till discharge from the ICU, assessed up to 1 year after the first day of admission.
  estimated Glomerular Filtration Rate (eGFR)
Renal function | Serum creatinine will be measured daily till discharge from the ICU, assessed up to 1 year after the first day of admission.
  serum creatinine
Need of renal replacement therapy | Need of renal replacement therapy during hospital admission will be determined at hospital discharge, assessed up to 1 year after the first day of admission.
  Yes or no
Medical Research Council score | Day 3, 5 and 7
  IC-acquired weakness
CAM-ICU score | Daily for 1 week
  Delirium
ICDSC score | Daily for 1 week
  Delirium
C-reactive protein | Daily for 1 week
  Inflammation
F2-isoprostanes | Daily from day 1 to 7
  Oxidative stress parameters
Oxidation-reduction potential | Day 1, 3 and 5
  Oxidative stress parameters
Antioxidant capacity | Day 1, 3 and 5
  Oxidative stress parameters
Vitamin C plasma concentrations | Daily from day 1 to 5

CONTACTS AND LOCATIONS:
Overall Officials: Angelique ME Spoelstra-de Man, Dr., Study Director — Amsterdam UMC, location VUmc
Locations (1):
- VU Medical Center, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grasner JT, Bottiger BW, Bossaert L; European Registry of Cardiac Arrest (EuReCa) ONE Steering Committee; EuReCa ONE Study Management Team. EuReCa ONE - ONE month - ONE Europe - ONE goal. Resuscitation. 2014 Oct;85(10):1307-8. doi: 10.1016/j.resuscitation.2014.08.001. Epub 2014 Aug 15. No abstract available. PMID 25132474
- [Background] Beesems JA, Stieglis R, Koster RW. Reanimatie buiten het ziekenhuis in Noord-Holland en twente: resultaten ARREST-onderzoek 2006-2011. 2012.
- [Background] Oudemans-van Straaten HM, Spoelstra-de Man AM, de Waard MC. Vitamin C revisited. Crit Care. 2014 Aug 6;18(4):460. doi: 10.1186/s13054-014-0460-x. PMID 25185110
- [Background] Stub D, Bernard S, Duffy SJ, Kaye DM. Post cardiac arrest syndrome: a review of therapeutic strategies. Circulation. 2011 Apr 5;123(13):1428-35. doi: 10.1161/CIRCULATIONAHA.110.988725. No abstract available. PMID 21464058
- [Background] Grooth HJ, Spoelstra-de Man AME, Oudemans-van Straaten HM. Early plasma Vitamin C concentration, organ dysfunction and ICU mortality. Intensive Care Medicine 2014; 40 (10 (Suppl 1)): S199.
- [Background] Levine M, Padayatty SJ, Espey MG. Vitamin C: a concentration-function approach yields pharmacology and therapeutic discoveries. Adv Nutr. 2011 Mar;2(2):78-88. doi: 10.3945/an.110.000109. Epub 2011 Mar 10. PMID 22332036
- [Background] Padayatty SJ, Sun H, Wang Y, Riordan HD, Hewitt SM, Katz A, Wesley RA, Levine M. Vitamin C pharmacokinetics: implications for oral and intravenous use. Ann Intern Med. 2004 Apr 6;140(7):533-7. doi: 10.7326/0003-4819-140-7-200404060-00010. PMID 15068981
- [Background] van Zanten AR, Sztark F, Kaisers UX, Zielmann S, Felbinger TW, Sablotzki AR, De Waele JJ, Timsit JF, Honing ML, Keh D, Vincent JL, Zazzo JF, Fijn HB, Petit L, Preiser JC, van Horssen PJ, Hofman Z. High-protein enteral nutrition enriched with immune-modulating nutrients vs standard high-protein enteral nutrition and nosocomial infections in the ICU: a randomized clinical trial. JAMA. 2014 Aug 6;312(5):514-24. doi: 10.1001/jama.2014.7698. PMID 25096691
- [Background] Baker TA, Milstien S, Katusic ZS. Effect of vitamin C on the availability of tetrahydrobiopterin in human endothelial cells. J Cardiovasc Pharmacol. 2001 Mar;37(3):333-8. doi: 10.1097/00005344-200103000-00012. PMID 11243424
- [Background] May JM, Qu ZC. Nitric oxide mediates tightening of the endothelial barrier by ascorbic acid. Biochem Biophys Res Commun. 2011 Jan 14;404(2):701-5. doi: 10.1016/j.bbrc.2010.12.046. Epub 2010 Dec 13. PMID 21156160
- [Background] Carr AC, Shaw GM, Fowler AA, Natarajan R. Ascorbate-dependent vasopressor synthesis: a rationale for vitamin C administration in severe sepsis and septic shock? Crit Care. 2015 Nov 27;19:418. doi: 10.1186/s13054-015-1131-2. PMID 26612352
- [Background] Jordan JE, Zhao ZQ, Vinten-Johansen J. The role of neutrophils in myocardial ischemia-reperfusion injury. Cardiovasc Res. 1999 Sep;43(4):860-78. doi: 10.1016/s0008-6363(99)00187-x. PMID 10615413
- [Background] Verma S, Fedak PW, Weisel RD, Butany J, Rao V, Maitland A, Li RK, Dhillon B, Yau TM. Fundamentals of reperfusion injury for the clinical cardiologist. Circulation. 2002 May 21;105(20):2332-6. doi: 10.1161/01.cir.0000016602.96363.36. No abstract available. PMID 12021216
- [Background] Huet O, Dupic L, Batteux F, Matar C, Conti M, Chereau C, Lemiale V, Harrois A, Mira JP, Vicaut E, Cariou A, Duranteau J. Postresuscitation syndrome: potential role of hydroxyl radical-induced endothelial cell damage. Crit Care Med. 2011 Jul;39(7):1712-20. doi: 10.1097/CCM.0b013e3182186d42. PMID 21494109
- [Background] Beale RJ, Sherry T, Lei K, Campbell-Stephen L, McCook J, Smith J, Venetz W, Alteheld B, Stehle P, Schneider H. Early enteral supplementation with key pharmaconutrients improves Sequential Organ Failure Assessment score in critically ill patients with sepsis: outcome of a randomized, controlled, double-blind trial. Crit Care Med. 2008 Jan;36(1):131-44. doi: 10.1097/01.CCM.0000297954.45251.A9. PMID 18007263
- [Background] Long CL, Maull KI, Krishnan RS, Laws HL, Geiger JW, Borghesi L, Franks W, Lawson TC, Sauberlich HE. Ascorbic acid dynamics in the seriously ill and injured. J Surg Res. 2003 Feb;109(2):144-8. doi: 10.1016/s0022-4804(02)00083-5. PMID 12643856
- [Background] Borrelli E, Roux-Lombard P, Grau GE, Girardin E, Ricou B, Dayer J, Suter PM. Plasma concentrations of cytokines, their soluble receptors, and antioxidant vitamins can predict the development of multiple organ failure in patients at risk. Crit Care Med. 1996 Mar;24(3):392-7. doi: 10.1097/00003246-199603000-00006. PMID 8625625
- [Background] Fowler AA 3rd, Syed AA, Knowlson S, Sculthorpe R, Farthing D, DeWilde C, Farthing CA, Larus TL, Martin E, Brophy DF, Gupta S; Medical Respiratory Intensive Care Unit Nursing; Fisher BJ, Natarajan R. Phase I safety trial of intravenous ascorbic acid in patients with severe sepsis. J Transl Med. 2014 Jan 31;12:32. doi: 10.1186/1479-5876-12-32. PMID 24484547
- [Background] Hume R, Weyers E, Rowan T, Reid DS, Hillis WS. Leucocyte ascorbic acid levels after acute myocardial infarction. Br Heart J. 1972 Mar;34(3):238-43. doi: 10.1136/hrt.34.3.238. No abstract available. PMID 5015020
- [Background] Tsai MS, Huang CH, Tsai CY, Chen HW, Cheng HJ, Hsu CY, Chang WT, Chen WJ. Combination of intravenous ascorbic acid administration and hypothermia after resuscitation improves myocardial function and survival in a ventricular fibrillation cardiac arrest model in the rat. Acad Emerg Med. 2014 Mar;21(3):257-65. doi: 10.1111/acem.12335. PMID 24628750
- [Background] Lloberas N, Torras J, Herrero-Fresneda I, Cruzado JM, Riera M, Hurtado I, Grinyo JM. Postischemic renal oxidative stress induces inflammatory response through PAF and oxidized phospholipids. Prevention by antioxidant treatment. FASEB J. 2002 Jun;16(8):908-10. doi: 10.1096/fj.01-0880fje. Epub 2002 Apr 23. PMID 12039876
- [Background] Seo MY, Lee SM. Protective effect of low dose of ascorbic acid on hepatobiliary function in hepatic ischemia/reperfusion in rats. J Hepatol. 2002 Jan;36(1):72-7. doi: 10.1016/s0168-8278(01)00236-7. PMID 11804667
- [Background] Ulug BT, Aksungar FB, Mete O, Tekeli F, Mutlu N, Calik B. The effect of vitamin C on ischemia reperfusion injury because of prolonged tourniquet application with reperfusion intervals. Ann Plast Surg. 2009 Feb;62(2):194-9. doi: 10.1097/SAP.0b013e318184ab74. PMID 19158533
- [Background] Nathens AB, Neff MJ, Jurkovich GJ, Klotz P, Farver K, Ruzinski JT, Radella F, Garcia I, Maier RV. Randomized, prospective trial of antioxidant supplementation in critically ill surgical patients. Ann Surg. 2002 Dec;236(6):814-22. doi: 10.1097/00000658-200212000-00014. PMID 12454520
- [Background] Collier BR, Giladi A, Dossett LA, Dyer L, Fleming SB, Cotton BA. Impact of high-dose antioxidants on outcomes in acutely injured patients. JPEN J Parenter Enteral Nutr. 2008 Jul-Aug;32(4):384-8. doi: 10.1177/0148607108319808. PMID 18596309
- [Background] Marik PE, Khangoora V, Rivera R, Hooper MH, Catravas J. Hydrocortisone, Vitamin C, and Thiamine for the Treatment of Severe Sepsis and Septic Shock: A Retrospective Before-After Study. Chest. 2017 Jun;151(6):1229-1238. doi: 10.1016/j.chest.2016.11.036. Epub 2016 Dec 6. PMID 27940189
- [Background] Berger MM, Soguel L, Shenkin A, Revelly JP, Pinget C, Baines M, Chiolero RL. Influence of early antioxidant supplements on clinical evolution and organ function in critically ill cardiac surgery, major trauma, and subarachnoid hemorrhage patients. Crit Care. 2008;12(4):R101. doi: 10.1186/cc6981. Epub 2008 Aug 7. PMID 18687132
- [Background] Heyland D, Muscedere J, Wischmeyer PE, Cook D, Jones G, Albert M, Elke G, Berger MM, Day AG; Canadian Critical Care Trials Group. A randomized trial of glutamine and antioxidants in critically ill patients. N Engl J Med. 2013 Apr 18;368(16):1489-97. doi: 10.1056/NEJMoa1212722. PMID 23594003
- [Background] Tanaka H, Matsuda T, Miyagantani Y, Yukioka T, Matsuda H, Shimazaki S. Reduction of resuscitation fluid volumes in severely burned patients using ascorbic acid administration: a randomized, prospective study. Arch Surg. 2000 Mar;135(3):326-31. doi: 10.1001/archsurg.135.3.326. PMID 10722036
- [Background] Hoffer LJ, Levine M, Assouline S, Melnychuk D, Padayatty SJ, Rosadiuk K, Rousseau C, Robitaille L, Miller WH Jr. Phase I clinical trial of i.v. ascorbic acid in advanced malignancy. Ann Oncol. 2008 Nov;19(11):1969-74. doi: 10.1093/annonc/mdn377. Epub 2008 Jun 9. PMID 18544557
- [Background] Stephenson CM, Levin RD, Spector T, Lis CG. Phase I clinical trial to evaluate the safety, tolerability, and pharmacokinetics of high-dose intravenous ascorbic acid in patients with advanced cancer. Cancer Chemother Pharmacol. 2013 Jul;72(1):139-46. doi: 10.1007/s00280-013-2179-9. Epub 2013 May 14. PMID 23670640
- [Background] Riordan HD, Casciari JJ, Gonzalez MJ, Riordan NH, Miranda-Massari JR, Taylor P, Jackson JA. A pilot clinical study of continuous intravenous ascorbate in terminal cancer patients. P R Health Sci J. 2005 Dec;24(4):269-76. PMID 16570523
- [Derived] Rozemeijer S, de Grooth HJ, Elbers PWG, Girbes ARJ, den Uil CA, Dubois EA, Wils EJ, Rettig TCD, van Zanten ARH, Vink R, van den Bogaard B, Bosman RJ, Oudemans-van Straaten HM, de Man AME. Early high-dose vitamin C in post-cardiac arrest syndrome (VITaCCA): study protocol for a randomized, double-blind, multi-center, placebo-controlled trial. Trials. 2021 Aug 18;22(1):546. doi: 10.1186/s13063-021-05483-3. PMID 34407846

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-03-05): https://cdn.clinicaltrials.gov/large-docs/62/NCT03509662/SAP_000.pdf